CLINICAL TRIAL: NCT06464120
Title: Investigating the Post-Activation Performance Enhancement Effects on Strength-trained Athletes Under Varied Loading Conditions: A Time-domain Features Perspective
Brief Title: Investigating the Post-Activation Performance Enhancement Effects on Skeletal Muscles Under Varied Loading Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Rong Wenchao, Study Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2024Y002
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Performance Enhancing Product Use
Keywords: Post-activation performance enhancement; strength training; take-off height; round reaction force; peak power

STUDY DESIGN:
Intervention Model Description: The experimental group was randomly assigned to receive strength training with increasing loads for post-activation enhancement intervention, while the control group received strength training with constant loads.
Masking Description: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental load training group (Experimental): This training plan is a single training，The load intensity of strength training for athletes :（5,4,3）RM×1 time ×1set for half squat jump
  Interventions: Other: Increasing load strength training
- Constant load training group (Experimental): This training plan is a single training，This training plan is a single training，Constant load of strength training for athletes :90%1RM×3 time ×1set for half squat jump
  Interventions: Other: Constant load strength training

INTERVENTIONS:
Other: Increasing load strength training — The Smith machine was used to intervene with athletes by employing an incremental load approach.
  Arms: Incremental load training group
Other: Constant load strength training — The Smith machine was used to intervene with athletes by employing a constant load approach.
  Arms: Constant load training group

SUMMARY:
With the advancement of sports science, Post-Activation Potentiation (PAP) has become a focal point of research, garnering significant attention for its underlying physiological mechanisms. Current studies suggest three primary mechanisms: 1) phosphorylation of myosin regulatory light chains (RLCs); 2) increased recruitment of high-threshold motor units; and 3) a reduction in sarcomere length heterogeneity within muscle fibers due to pre-stimulation (Liu & Li, 2017). These mechanisms collectively contribute to an effect known as Post-Activation Performance Enhancement (PAPE), which significantly enhances muscle strength and explosiveness shortly after activation (Blazevich & Babault, 2019).

During the activation process of motor units with increasing loads, low-threshold motor units are recruited first, followed by high-threshold motor units. As the load increases, the root mean square (RMS) value increases linearly, further promoting the overlap of motor unit potentials and the rise in RMS values. This overlap in activation timing among adjacent motor units results in greater overall muscle force output (Liu, 2008; Tian, 2009). The significance of this lies in the fact that as the degree of muscle activation increases, especially under incremental loads, the muscle's ability to adapt to subsequent strength or explosive tasks may be enhanced.

In competitive sports, optimizing the relationship between warm-up and performance is crucial. Research indicates that the duration of PAPE varies with individual differences, training type, intensity, and recovery intervals. The characteristics of the PAPE effect also differ. Additionally, following constant loads, the enhancement and decay rates of performance in PAPE show varying rates at different times, and these rates do not exhibit a symmetrical linear change in absolute value (Liang, M 2020; Guo, W et al. 2018; Liu, R and Li, Q. 2017). The competition pace in sports demands precise modulation of performance enhancement rates after activation, and athletes can leverage these characteristics by selecting appropriate loading forms to trigger PAPE at critical moments in competition. To explore the enhancement or decay rates of performance over different time domains, our research team designed a protocol consisting of incremental loads.

DETAILED DESCRIPTION:
First, participants underwent a squat 1-RM test using the NSCA testing protocol. The induction exercise was barbell-loaded squats. In the constant load group, the stimulation intensity was set at 90% of the 1-RM, with one set of four repetitions of barbell half-squat jumps . In the incremental load group, the stimulation intensities were set at 5RM, 4RM, 3RM, and 2RM, with one set of one repetition of barbell half-squat jumps for each load intensity. Both the 1-RM test and squat induction exercises were conducted using a Smith machine, and protective personnel were present on both sides. The testing movement involved static half-squat jumps that aimed to enhance the stability of the test and reduce interference from arm swinging. The static half-squat jump required participants to stand with their feet shoulder-width apart on the force plate, hands on hips, and knees flexed to a semi-movement range, and they had to maintain the position for one to two seconds. Following this, participants exerted maximal effort to jump upward (with no visually noticeable downward squatting during takeoff) before naturally descending and maintaining the position for another one to two seconds. Throughout the entire process, both feet were to remain within the force plate area.

Experimental procedure The participants began with a 10-minute slow jog and dynamic lower-limb stretches. As a baseline, the participants' dynamic data for unloaded static half-squat jumps were collected after a 5-minute rest. Following another 5-minute rest, the constant load group underwent one set of four half-squat jump inductions at an intensity of 90% 1-RM. The incremental load group underwent inductions at each load intensity, with one set of barbell half-squat jump exercises for each intensity. The participants received verbal cues and encouragement for each repetition. Dynamic data for static half-squat jumps were collected at 15 seconds, 3 minutes, 6 minutes, 9 minutes, and 12 minutes after the end of each exercise session. At each time point, two valid repetitions were collected, with verbal cues and encouragement provided to the participants for each repetition. Each set of two half-squat jumps did not exceed 10 seconds. The interval between static half-squat jump testing and 1-RM testing was greater than 48 hours .

ELIGIBILITY:
Inclusion Criteria:

(1) Voluntary participation in the research study with prior experience in weighted deep squat exercises; (2) No intake of caffeine within 3 hours before testing and no high-intensity resistance exercises for the lower limbs within the past 24 hours; (3) No lower limb joint injuries (open or closed), no cardiovascular diseases, no skin allergies, and no symptoms of hernia in the last 12 months; (4) Maintenance of regular diet and sleep patterns during the study, and exclusion from any additional strength training activities apart from normal daily life.

Exclusion Criteria:

(1) Individuals with a history of lower limb joint injuries; (2) Individuals with cardiovascular diseases, skin allergies, hernia, or any other contraindications; (3) Individuals unwilling to participate in the experiment.

Ages: 19 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Ground reaction force | 30 seconds, 3 minutes, 6 minutes, 9 minutes, 12 minutes after intervention and before intervention
  The ground reaction force of the lower limbs during the half squat jump was measured by the force platform.
Peak Power | 30 seconds, 3 minutes, 6 minutes, 9 minutes, 12 minutes after intervention and before intervention
  Athletes measured the peak power of the lower limbs in the half squat jump using a force platform
Height | 30 seconds, 3 minutes, 6 minutes, 9 minutes, 12 minutes after intervention and before intervention
  The athlete uses a 3D motion capture device to measure the height of the highest point of the half squat jump

CONTACTS AND LOCATIONS:
Overall Officials: wenchao Rong, phd, Principal Investigator — University Putra Malaysia
Locations (1):
- RongWenchao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No
I won't share it, until I published this paper